CLINICAL TRIAL: NCT07295925
Title: Prospective Evaluation of Clinical, Laboratory and Operative Predictors of Postoperative Fever and Sepsis After Retrograde Intrarenal Surgery (RIRS)
Brief Title: Risk Factors for Postoperative Fever and Sepsis Following Retrograde Intrarenal Surgery
Acronym: SARIS
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Emre Can Akınsal, Emre Can Akınsal Assoc. Prof., TC Erciyes University
Other Study IDs: SEPSIS_AFTER_RIRS_26
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Urolithiasis
Keywords: RIRS; Sepsis; Urolithiasis; Endourology; Retrograde Intrarenal Surgery; Postoperative Fever; Postoperative Sepsis; Ureteroscopy
MeSH Terms: conditions — Urolithiasis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RIRS Patient Group: Patients undergoing retrograde intrarenal surgery (RIRS) for urinary stone disease who are prospectively followed to identify clinical, laboratory and operative predictors of postoperative fever and sepsis

SUMMARY:
This prospective clinical study aims to evaluate preoperative, intraoperative, and postoperative characteristics of patients undergoing retrograde intrarenal surgery (RIRS) for urinary stone disease. A total of approximately 250 patients will be assessed to identify clinical, laboratory, and operative factors associated with postoperative fever and sepsis. By systematically collecting and analyzing perioperative data, the study seeks to determine independent predictors that may support improved risk stratification and patient safety in endourological practice.

DETAILED DESCRIPTION:
Urinary stone disease is a common global health problem with an increasing incidence and significant clinical and economic burden. Retrograde intrarenal surgery (RIRS) has become a widely accepted, minimally invasive, and effective treatment option for renal and proximal ureteral stones. Advances in flexible ureteroscope design, laser technologies, and endourological instrumentation have further improved the safety, efficiency, and applicability of RIRS. As a result, there has been a marked increase in the preference for RIRS among urologists in recent years.

Despite its advantages, RIRS is associated with complication rates reported between 9% and 25%. Postoperative fever and urinary tract infection are the most frequently observed complications and may progress to sepsis, which represents a potentially life-threatening condition in patients with urinary stone disease. These infectious events remain a concern even when appropriate antibiotic prophylaxis and aseptic surgical principles are applied. Identifying risk factors that may predict postoperative infection and sepsis is therefore essential for improving perioperative decision-making and patient safety.

Previous studies have suggested potential associations between operative characteristics, preoperative bacteriuria, patient-related comorbidities, and postoperative infectious outcomes; however, most available evidence originates from retrospective analyses with limited variables. There remains a need for prospective, systematically collected data evaluating a broad set of perioperative clinical and laboratory parameters to better define predictive factors.

This prospective patient registry study aims to evaluate comprehensive perioperative variables to identify predictors of postoperative urinary tract infection and sepsis following RIRS. Parameters to be assessed include operative time, stone burden, intraoperative irrigation characteristics, perioperative cultures, and a detailed panel of inflammatory biomarkers such as C-reactive protein, procalcitonin, albumin, fibrinogen, and D-dimer. The study will also record the onset, duration, and severity of postoperative fever, together with other clinical findings relevant to infectious complications. Through this structured approach, the study seeks to determine independent risk factors that may assist clinicians in predicting, preventing, and managing postoperative infection and sepsis in patients undergoing RIRS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients scheduled to undergo retrograde intrarenal surgery (RIRS) for the treatment of renal or ureteral stones.
* Completion of routine preoperative and postoperative clinical assessments required for RIRS.
* Ability to provide informed consent.

Exclusion Criteria:

* Terminal-stage malignancy.
* Bleeding diathesis or known immunodeficiency.
* Active infectious condition at the time of surgery.
* Patients deemed unsuitable for anesthesia or surgery by the Department of Anesthesiology.
* Pregnancy.
* Contraindications to RIRS or inability to complete required perioperative evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing retrograde intrarenal surgery (RIRS) for the treatment of renal or ureteral stones at Erciyes University Hospital. All participants are evaluated using standard preoperative laboratory tests, imaging studies, and perioperative clinical assessments. Patients included in this registry represent a typical endourological population treated with RIRS in routine clinical practice. Individuals with active infections at the time of surgery, contraindications to surgery, or conditions preventing informed consent are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Postoperative Sepsis | Within 72 hours after surgery
  Postoperative sepsis will be defined according to Sepsis-3 criteria, based on suspected or confirmed infection and an increase of ≥ 2 points in the Sequential Organ Failure Assessment (SOFA) score within 72 hours after retrograde intrarenal surgery (RIRS).

SECONDARY OUTCOMES:
Number of Participants With Postoperative Fever | Within 72 hours after surgery
  Postoperative fever will be defined as a body temperature ≥38ºC recorded at least twice within 72 hours after retrograde intrarenal surgery (RIRS).
Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) | First 24 hours after surgery
  SIRS will be defined according to standard clinical criteria, including abnormalities in body temperature, heart rate, respiratory rate and leukocyte count after retrograde intrarenal surgery (RIRS).
Number of Participants With Positive Postoperative Urine Culture | Within 72 hours
  Growth of ≥10⁵ CFU/mL of a single organism in a postoperative urine culture.
Number of Participants with Positive Postoperative Blood Culture | Within 72 hours
  Detection of pathogenic microorganisms from blood samples obtained in the postoperative period.
Number of Participants With Positive Stone Culture | Up to 72 hours after surgery
  Presence of bacterial growth in stone culture obtained during retrograde intrarenal surgery (RIRS), defined as any clinically significant pathogen isolated from stone fragments
Length of Hospital Stay (days) | From the date of surgery until hospital discharge, assessed up to 30 days postoperatively.
  Length of hospital stay will be defined as the number of days from the date of surgery to the date of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Emre C. Akınsal, Assoc. Prof., Principal Investigator — Erciyes University Faculty of Medicine, Department of Urology; Emre C. Akınsal, Assoc. Prof., Study Chair — Erciyes University Faculty of Medicine, Department of Urology
Locations (1):
- Erciyes University Faculty of Medicine, Department of Urology, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No